CLINICAL TRIAL: NCT03029312
Title: Whole Body Vibration as an Osteogenic Treatment for Children With Osteogenesis Imperfecta With Limited Mobility: A Randomised Controlled Pilot Trial
Brief Title: Whole Body Vibration Training in Children With Osteogenesis Imperfecta and Limited Mobility
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Birmingham Women's and Children's NHS Foundation Trust (Other)
Collaborators: Royal Manchester Children' s Hospital, Manchester (Unknown); University of Sheffield (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11/WM/0275
Record Dates: First submitted 2017-01-19; First posted 2017-01-24 (Estimated); Last update posted 2017-01-24 (Estimated); Status verified 2017-01

CONDITIONS: Osteogenesis Imperfecta
Keywords: whole body vibration; Muscle function; Physical activity; bone density
MeSH Terms: conditions — Osteogenesis Imperfecta; Motor Activity

STUDY DESIGN:
Intervention Model Description: Paired randomized controlled study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | US Export: No

ARMS (2):
- Whole Body Vibration (Experimental): Twice daily WBVT at home using the Galileo M device, 3x3 min, with 3 minute breaks (total daily WBVT 18 min) for 5 months. Children stand upright on the device, with knees bent (10-45 degrees, semi-squat or squat position). A schedule of increasing intensity of vibration exercise was used over time, allowing some adjustment to the patient's physical capability. Amplitude 1 was used for the first 2 weeks, then increased to amplitude 2 and further increased up to amplitude 3, if individually possible, always using frequencies between 20-25Hz. Children also perform exercises on the platform, including shifting their weight from one side to the other, increase/decrease their knee and hip angle, weight shift with trunk rotation, and alternate flexion and extension of knees.
  Interventions: Device: Galileo M
- Regular Care (No Intervention): Regular Care, including physiotherapy for 5 months

INTERVENTIONS:
Device: Galileo M — Motorized board producing side-to-side alternating vertical sinusoidal (rotational) vibrations around a fulcrum in the mid-section of the plate. The vibration frequency can be selected by the user who stands on the board with both feet, wearing shoes. The peak-to-peak displacement to which the feet are exposed increases with the distance of the feet from the centre line of the vibrating board. Three positions marked 1, 2 and 3 are indicated on the vibrating board, corresponding to peak-to-peak displacements of 2, 4, and 6mm. The peak acceleration exerted by vibration exercise increases with higher frequencies and higher amplitudes.
  Other Names: Vibraflex
  Arms: Whole Body Vibration

SUMMARY:
Children with osteogenesis imperfecta (OI) have impaired bone strength, fractures, weak muscles and limited mobility. Mild to moderate forms of OI (type 1 and 4) may benefit from muscle training that leads to secondary improvement in bone strength (osteogenic treatment). Recent studies in children with cerebral palsy but also OI suggest that Whole Body Vibration Training (WBVT) improves mobility and also bone strength. No randomized controlled trials exist in OI children. This randomized controlled pilot study assesses the effect of 5 months WBVT (2 x 9min/day) on muscle function, mobility, bone structure and density. 24 children >5 years with OI type 1 and 4 with limited mobility (CHAQ Score ≥0.13) will be randomized into a WBVT group and a control group matched by gender and pubertal stage. Main outcome measure is the change in tibial volumetric BMD, secondary outcomes include a variety of bone, mobility and dynamic muscle function variables.

DETAILED DESCRIPTION:
Osteogenesis imperfecta (OI) is a bone fragility disorder with impaired bone strength, fractures, weak muscles and limited mobility. Mild to moderate forms of OI (type 1 and 4) may not require bisphosphonate therapy but would benefit from muscle training that leads to secondary improvement in bone strength (osteogenic treatment). The mechanostat theory states that bone adapts its strength to mechanical forces mostly imposed by muscle. According to this widely accepted theory, any treatment that strengthens muscle should also strengthen bones. Whole body vibration therapy (WBVT) with side-alternating platforms (Galileo™) uses the body's neuromotor reflex system to train muscles. Recent studies in children with cerebral palsy but also OI suggest that WBVT improves mobility and also bone strength. No randomized controlled trials exist in OI children.

This randomized controlled study assesses the effect of 5 months whole body vibration training (2 x 9min/day) on muscle strength, motor function, bone structure and density. 24 children >5 years with OI type 1 and 4 with limited mobility (CHAQ Score ≥0.13) will be randomized into a WBVT group and a control group matched by gender and pubertal stage. Children with OI will be recruited from specialist clinics in Birmingham, Manchester and Sheffield, as well as via advertisement on the Brittle Bone Society's homepage. Patients will be equipped with side-alternating vibration platforms for home use and train with increasing intensity. Outcome measures are tested pre- and post 5-months intervention. Dynamic muscle function is measured by mechanography (jumping force plates) and mobility by CHAQ questionnaire and a six-minute walk test. Changes in bone structure and density are assessed by DXA and peripheral QCT of the tibia.

ELIGIBILITY:
Inclusion Criteria:

Patients with mild OI (type 1 and 4; >5y of age) who need to be at least partly ambulant and have a CHAQ score of greater than 0.13, constituting at least mild disability. Minimum requirement is the ability to rise from a chair.

Informed consent is required from the participant and/or parent/guardian.

-

Exclusion Criteria:

* On bisphosphonate treatment for less than 2years (since mobility usually improves during the initial phase treatment).
* Finished bisphosphonate therapy less than 6 months ago
* Recent lower limb fracture <3months ago, or upper limb fracture which is still in plaster.
* Heart or lung disease, use of steroids (oral, systemic, topical or inhaled, for more than 3 weeks in the last 12 months) or any other bone-active treatment.

Ages: 5 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes — 12 boys, 12 girls
Enrollment: 24 (Actual)
Dates: Start 2012-01-17 (Actual); Primary Completion 2015-11-18 (Actual); Study Completion 2016-01-18 (Actual)

PRIMARY OUTCOMES:
Does WBVT increase bone density at the distal tibia | 5 months
  Trabecular volumetric BMD measured at the distal tibia (4% of tibia length)

SECONDARY OUTCOMES:
Does WBVT result in an increase in dynamic muscle function | 5 months
  Jumping Mechanography (single 2-leg jump, multiple one leg hop, chair and heel rise test)
Does WBVT result in an increase in muscle mass | 5 months
  Muscle mass measured by DXA
Does WBVT result in an increase in density | 5 months
  Bone density measured by DXA
Does WBVT result in an increase in density of the tibia | 5 months
  Bone density measured by pQCT
Does WBVT result in an increase in bone geometry | 5 months
  Bone size measured by pQCT
Does WBVT result in an increase in 6-minute walking distance | 5 months
  six minute walk tests
Does WBVT result in improved disability | 5 months
  CHAQ disability score
Does WBVT result in improved balance | 5 months
  Balance (sway area measured by mechanography)

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang Högler, MD PD, Principal Investigator — Birmingham Children's Hospital
Locations (1):
- Birmingham Children's Hospital, Birmingham, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Anonymised data available on request, subject to Ethical and R&D guidelines

REFERENCES:
- [Derived] Hogler W, Scott J, Bishop N, Arundel P, Nightingale P, Mughal MZ, Padidela R, Shaw N, Crabtree N. The Effect of Whole Body Vibration Training on Bone and Muscle Function in Children With Osteogenesis Imperfecta. J Clin Endocrinol Metab. 2017 Aug 1;102(8):2734-2743. doi: 10.1210/jc.2017-00275. PMID 28472303